CLINICAL TRIAL: NCT04837872
Title: Static Progressive Splinting in the Management of Knee Stiffness Following Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Panorama Orthopedics & Spine Center (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-0241
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: static progressive splinting; manual therapy; physical therapy; rehabilitation; arthrofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Physical Therapy (MPT) (Experimental): The multimodal physical therapy (MPT) program consisted of manual therapy, therapeutic exercise, and utilization of a static progressive splint (Joint Active Systems SPS Knee, Effingham, IL). Although the primary focus of this study was on improving knee flexion ROM, two protocols were developed: one to improve flexion deficits and one to improve extension deficits. Participants in the MPT group received physical therapy 2x per week for 4 weeks. They were instructed to use the static progressive splint(s) 3x per day for 30 minute sessions (90 minutes total per day) for each splint (e.g., 90 minutes for flexion splint, 90 minutes for extension splint).
  Interventions: Other: Multimodal Physical Therapy (MPT)

INTERVENTIONS:
Other: Multimodal Physical Therapy (MPT) — Individualized physical therapy and static progressive splint (flexion with or without extension splint).

SUMMARY:
The purpose of this study is to determine the feasibility and initial efficacy of static progressive splinting for individuals presenting with knee stiffness following total knee arthroplasty (TKA). Data from this trial will be utilized in a NIH grant application for a larger randomized controlled trial directly comparing static progressive splinting to manipulation under anesthesia (MUA) which is the current standard of care for knee stiffness after TKA.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the standard of care to manage the pain and disability associated with end-stage knee osteoarthritis, with more than 700,000 TKA surgeries performed annually in the United States. Knee stiffness, commonly caused by arthrofibrosis, is an infrequent, but debilitating complication of TKA, with an incidence upwards of 5% postoperatively. As a predominant failure mechanism, knee stiffness accounts for 28% of hospital readmissions due to surgical complications within 90 days of discharge, and 10% of all revisions within 5 years of initial surgery within the United States. With the incidence of TKA projected to reach 3.5 million by 2030, the growing cohort of TKA patients with postoperative knee stiffness provides an important target for research.

Several treatments for knee stiffness have been described including static progressive splinting and manipulation under anesthesia (MUA). To date, no studies have compared the use of static progressive splinting in the early management of individuals presenting with knee stiffness after TKA to more commonly utilized surgical procedures such as MUA. Witvrouw and colleagues compared a computer-controlled passive motion device to MUA for individuals with knee stiffness after TKA and found that stretching device had similar outcomes to MUA in terms of range of motion (ROM) and self-reported pain, stiffness and function. A key limitation of this study is that the computer-controlled motion device is not commercially available and therefore translation of this technology into practice is unlikely. However, this study does demonstrate that conservative stretching techniques may be as efficacious as costlier surgical techniques as well as may cause fewer adverse events such as quadriceps tendon rupture and fractures. Only one study to date has examined the utilization of static progressive splinting after TKA. In this study, they enrolled patients who had already failed MUA and conservative physical therapy management strategies. They found that the average ROM increase for patients was 25° as well as 92% of patients were satisfied with the results and no complications occurred with use of the device. Key limitations to this study are the lack of a comparison group as well as static progressive splinting was utilized after MUA had already failed. It is unknown how individuals would respond to this treatment compared to MUA.

Therefore, the purpose of our study is to determine the feasibility and initial efficacy of static progressive splinting for individuals presenting with knee stiffness following TKA within the current surgical practice of Dr. Jared Foran at Panorama Orthopedics & Spine Center. Data from this trial will be utilized in a NIH grant application for a larger randomized controlled trial directly comparing static progressive splinting to MUA which is the current standard of care for knee stiffness after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Undergone a unilateral primary Total Knee Arthroplasty (TKA) for end-stage osteoarthritis
* Knee stiffness in the first 6 weeks post-operative defined as knee flexion < 100 degrees

Exclusion Criteria:

* Preoperative knee range of motion less than 15-110 degrees
* Intraoperative (closed) range of motion < 0-120 degrees
* Radiographic signs of heterotopic ossification
* Misaligned components or component-related failures of knee prosthesis that could be responsible for difficulties with motion
* Signs and symptoms consistent with joint infection
* Signs and symptoms consistent with complex regional pain syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 4 weeks
  Passive knee flexion and extension measured with goniometry

SECONDARY OUTCOMES:
Adherence to Splint Use | 4 weeks
  Adherence to splint use was tracked with a log completed by participants; they were instructed to place a checkmark for each day they used the JAS splint per protocol (30-minute sessions, 3 times daily). Adherence was calculated as days of splint use completed divided by days of splint use prescribed; a priori adherence levels were considered acceptable if the mean was ≥ 80 percent.
Satisfaction with Splint | 4 weeks
  Satisfaction was assessed with a 7-point Likert scale ranging from 1 "extremely dissatisfied" to 7 "extremely satisfied". Participants responded based on the following instruction: please rate your satisfaction with your knee splint on the scale. A priori satisfaction was considered acceptable if the median score was ≥ 4 ("somewhat satisfied" or higher).
Safety of splint use: adverse events | 4 weeks
  Count and description of adverse events related to splint use

CONTACTS AND LOCATIONS:
Locations (1):
- Panorama Orthopedics & Spine Center, Golden, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yercan HS, Sugun TS, Bussiere C, Ait Si Selmi T, Davies A, Neyret P. Stiffness after total knee arthroplasty: prevalence, management and outcomes. Knee. 2006 Mar;13(2):111-7. doi: 10.1016/j.knee.2005.10.001. Epub 2006 Feb 20. PMID 16490357
- [Background] Schroer WC, Berend KR, Lombardi AV, Barnes CL, Bolognesi MP, Berend ME, Ritter MA, Nunley RM. Why are total knees failing today? Etiology of total knee revision in 2010 and 2011. J Arthroplasty. 2013 Sep;28(8 Suppl):116-9. doi: 10.1016/j.arth.2013.04.056. Epub 2013 Aug 15. PMID 23954423
- [Background] Schairer WW, Vail TP, Bozic KJ. What are the rates and causes of hospital readmission after total knee arthroplasty? Clin Orthop Relat Res. 2014 Jan;472(1):181-7. doi: 10.1007/s11999-013-3030-7. PMID 23645339
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Bonutti PM, Marulanda GA, McGrath MS, Mont MA, Zywiel MG. Static progressive stretch improves range of motion in arthrofibrosis following total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2010 Feb;18(2):194-9. doi: 10.1007/s00167-009-0947-1. Epub 2009 Oct 14. PMID 19826784
- [Background] Manrique J, Gomez MM, Parvizi J. Stiffness after total knee arthroplasty. J Knee Surg. 2015 Apr;28(2):119-26. doi: 10.1055/s-0034-1396079. Epub 2014 Dec 16. PMID 25513992
- [Background] Witvrouw E, Bellemans J, Victor J. Manipulation under anaesthesia versus low stretch device in poor range of motion after TKA. Knee Surg Sports Traumatol Arthrosc. 2013 Dec;21(12):2751-8. doi: 10.1007/s00167-012-2152-x. Epub 2012 Aug 3. PMID 22864680
- [Derived] Rauzi MR, Foran JRH, Bade MJ. Multimodal conservative management of arthrofibrosis after total knee arthroplasty compared to manipulation under anesthesia: a feasibility study with retrospective cohort comparison. Pilot Feasibility Stud. 2022 Mar 25;8(1):71. doi: 10.1186/s40814-022-01026-y. PMID 35337388
- See also: Most Frequent Operating Room Procedures Performed in U.S. Hospitals, 2003-2012 — http://www.hcup-us.ahrq.gov/reports/statbriefs/sb186-Operating-Room-Procedures-United-States-2012.jsp